CLINICAL TRIAL: NCT07319156
Title: Assessment of Upper Extremity Proprioception in Patients With Cervical Radiculopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MarmaraU-FTR-FBA-02
Record Dates: First submitted 2025-12-01; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cervical Radiculopathy; Proprioception; Cervical Disc Herniation; Proprioception Reaching Test; Pro-reach; Upper Extremity
Keywords: cervical radiculopathy; proprioception; cervical disc herniation; proprioception reaching test; pro-reach; upper extremity
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Cervical Radiculopathy: Patients aged 18-65 years who were diagnosed with cervical radiculopathy based on history, physical examination, and clinical evaluation
- Healty Participants: Healthy volunteers matched to the cervical radiculopathy group in terms of age, sex, and BMI.

SUMMARY:
There is no study in the current literature that systematically investigates the extent of upper-extremity proprioceptive impairment in patients with radicular neuropathic symptoms secondary to cervical disc herniation, nor its association with clinical findings. Although existing reviews emphasize proprioceptive deficits in populations with neck pain or cervical spondylosis, no studies specifically address the subgroup of cervical disc-related radiculopathy. This gap in knowledge hinders the integration of proprioceptive assessments with upper-extremity functional outcome measures in diagnostic and rehabilitative processes, suggesting a need for more specific data to guide sensory-motor training approaches. The primary aim of the present study is to assess upper-extremity proprioception in patients with cervical radiculopathy by comparing them with a healthy control group. The secondary aim is to examine the relationship between upper-extremity proprioception and clinical outcomes, including parameters such as pain and functional status.

DETAILED DESCRIPTION:
Cervical radicular pain is a neuropathic pain syndrome characterized by dermatomal distribution resulting from irritation of the cervical spinal nerve roots. The most common underlying causes are cervical disc herniation and cervical spinal stenosis. Motor, sensory, or reflex disturbances may accompany the condition, and it is most frequently observed in individuals aged 50-54 years.

Proprioception is a sensorimotor function that enables the perception of joint position and movement through the processing of afferent inputs originating from joints, muscles, and tendons within the central nervous system. Proprioceptive inputs from the cervical spine integrate with visual and vestibular information to play a critical role in head-trunk orientation, postural control, and upper-extremity movement coordination.

Although there is currently no gold-standard method for assessing active joint position sense-the quantifiable component of proprioception-tools such as manual and digital goniometers, inclinometers, and laser pointers are commonly used. However, these techniques measure joint position sense in a single plane and typically at a single joint. Recent studies, however, support the use of assessment methods that capture multisensory spatial representation of the entire limb and reflect the complexity of daily functional movements by incorporating multiplanar and multi-joint measurements. The PRO-Reach method developed by Ager et al. enables such multi-planar and multi-joint assessment without requiring computerized interfaces or robotic devices.

Numerous studies have demonstrated impaired cervical proprioception in cervicogenic conditions such as chronic neck pain and cervical spondylosis. The aim of the present study is to investigate the extent of upper-extremity proprioceptive impairment in patients with cervical radiculopathy. Cervical muscle fatigue or alterations in cervical sensory input may reduce the accuracy of upper-extremity joint positioning, thereby negatively affecting upper-extremity proprioception

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years of age
* Presence of radicular pain diagnosed through clinical examination and cervical -MRI imaging Patients with cervical MRI findings demonstrating cervical disc herniation at least at one level consistent with their symptoms
* Willingness to participate in the study

Exclusion Criteria:

* History of cervical physical therapy within the past year
* Symptoms or diagnosis of upper-extremity entrapment neuropathy
* Patients with documented vitamin B12 or vitamin D deficiency within the last 2 years in available medical records
* History of cervical surgery or cervical trauma
* History of upper-extremity surgery or trauma
* Individuals with intellectual disability
* Presence of major psychiatric comorbidity
* Diagnosis of polyneuropathy
* Diagnosis of Diabetes Mellitus
* Diagnosis of fibromyalgia
* Use of medications that may impair proprioception
* Pregnancy
* Refusal to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years who are diagnosed with cervical radiculopathy based on history, physical examination, and clinical evaluation will be assessed according to the inclusion and exclusion criteria. Two groups will be formed: the cervical radiculopathy group and a healthy volunteer group matched for age, sex, and BMI.
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The Upper Limb Proprioception Reaching Test (PRO-Reach) | Baseline
  PRO-Reach is a 90 × 110 cm plastic poster mounted on the wall using bilateral magnetic strips. Round stickers with a diameter of 0.6 cm, manually numbered (1-3), are used to mark the three free-reach attempts for each target. Seven targets are used and are named according to the movement direction of the dominant limb: the left side of the poster represents the dominant side for left-handed participants, while the right side corresponds to non-dominant (ND) cross-body movements. The opposite applies to right-handed participants. The targets are labeled as follows: superior (S), superior-lateral dominant (SLD) and non-dominant (SLND), lateral-dominant (LD) and non-dominant (LND), and inferior-lateral dominant (ILD) and non-dominant (ILND). The (S) target is used for evaluation in participants without limb dominance. The (S) target is also used for the three familiarization trials (three memorization and reposition attempts). The purpose is to "assess the ability to reproduce movements

SECONDARY OUTCOMES:
The Numeric Rating Scale (NRS) | Baseline
  The Numeric Rating Scale (NRS) is a unidimensional, self-reported measure of pain intensity that is widely used in both clinical practice and research, including studies involving patients with chronic pain. On this scale, patients rate their current level of pain on an 11-point numeric range from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable." Higher scores indicate greater pain intensity.
DN-4 Quastionnaire | Baseline
  The DN-4 (Douleur Neuropathique en 4 Questions) is a brief and reliable screening questionnaire used to determine whether a patient's pain is of neuropathic origin. It consists of a total of 10 items. Its name, DN-4, derives from the fact that it includes 4 main sections. Seven of the questions relate to patient-reported sensory symptoms, while three are based on clinical examination findings. Each "yes" response scores 1 point, yielding a total score ranging from 0 to 10. A score above 4 indicates a high likelihood of neuropathic pain.
SHORT FORM-12 | Baseline
  The Short Form-12 (SF-12) is a health-related quality of life assessment tool that summarizes an individual's physical and mental health status through 12 items. It is a shortened version of the SF-36 questionnaire and measures eight health domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The SF-12 produces two composite scores - the Physical Component Summary (PCS) and the Mental Component Summary (MCS) - which are standardized to a mean of 50 and a standard deviation of 10 in the general population. Higher scores indicate better health status and quality of life.
Handgrip Strength Test(Jamar Hand Dynamometer) | Baseline
  The Jamar hand dynamometer is a hydraulic measurement device used to assess hand grip strength in an objective and reproducible manner. It is considered the gold standard in musculoskeletal research, rehabilitation, neurological evaluation, and work capacity assessments. The patient is seated with back support, the shoulder in a neutral position, the elbow flexed at 90°, and the forearm in a neutral position. The dynamometer is placed in the patient's hand, and they are instructed to "squeeze maximally." Typically, three trials are performed for each hand, and either the highest value or the mean value is used. Measurements are generally recorded in kilograms (kg) or pounds (lb). Higher scores indicate greater grip strength, whereas lower scores suggest reduced muscle strength and may reflect sarcopenia, as well as potential neurological or musculoskeletal functional impairment.
Quick Disabilities of the Arm, Shoulder and Hand Questionnaire (QuickDASH) | Baseline
  The QuickDASH (Quick Disabilities of the Arm, Shoulder and Hand) is a brief and practical self-report questionnaire used to assess functional impairment and symptom severity of the upper extremity. It is the shortened version of the full DASH questionnaire and is widely preferred in clinical practice. The scale consists of 11 items that evaluate functional limitations and symptoms such as pain in the hand, arm, and shoulder regions. Patients respond based on their condition over the past week. Each item is scored from 1 to 5, and the final score is calculated on a 0-100 scale. A score of 0 indicates no disability related to the upper extremity, whereas higher scores reflect greater levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma B Akdağ, Research Assistant, Principal Investigator — Marmara University Faculty of Medicine ,Marmara University, Department of Physical Medicine and Rehabilitation; Osman H Gündüz, Professor, Study Director — Algology Division, Department of Physical Medicine and Rehabilitation, Marmara University Faculty of Medicine; Serdar Kokar, Associate Professor, Study Director — Algology Division, Department of Physical Medicine and Rehabilitation, Marmara University Faculty of Medicine; Savaş Şencan, Associate Professor, Study Director — Algology Division, Department of Physical Medicine and Rehabilitation, Marmara University Faculty of Medicine; Gökçenur Yalçın, Medical specialist, Study Director — Marmara University Faculty of Medicine ,Marmara University, Department of Physical Medicine and Rehabilitation
Locations (1):
- Marmara University Faculty of Medicine, Pendik Training and Research Hospital, Algology Department, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No